CLINICAL TRIAL: NCT01365988
Title: Neural Correlates of Risk-Taking in Urban Adolescents
Brief Title: Neutral Correlates of Risk-taking in Adolescents Exposed to Drugs Prenatally
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911468; 11-DA-N468
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-02-26

CONDITIONS: Exposure
Keywords: fMRI; Risk-Taking; Decision-Making; Memory; Resting-State Functional Connectivity
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Objective- To use fMRI to compare brain activity at rest and during memory and decision making tasks in normal children and in children exposed in utero to drugs of abuse.

Study population- All participants will be 14-20 year-olds enrolled in an ongoing longitudinal follow up study of children exposed to drugs of abuse in utero funded by NIH. A subgroup of this study cohort will be invited to participate based on added criteria needed for scanning studies, such as absence of metal in the body, no significant CNS disease, and ability to tolerate the scanning environment.

Design- Participants will undergo fMRI scans while performing a memory task, a decision making task and at rest. Data from participants in the current study may be combined with those from a previous study (NIDA protocol 417) which now reside in our repository protocol, 8002 and NIDA protocol 455.

Outcome measures- The primary outcome measures will be the difference in BOLD fMRI activation between drug-exposed participants and those without prenatal exposure to drugs of abuse.

DETAILED DESCRIPTION:
Objective- To use fMRI to compare brain activity at rest and during memory and decision making tasks in normal children and in children exposed in utero to drugs of abuse.

Study population- All participants will be 14-20 year-olds enrolled in an ongoing longitudinal follow up study of children exposed to drugs of abuse in utero funded by NIH. A subgroup of this study cohort will be invited to participate based on added criteria needed for scanning studies, such as absence of metal in the body, no significant CNS disease, and ability to tolerate the scanning environment.

Design- Participants will undergo fMRI scans while performing a memory task, a decision making task and at rest. Data from participants in the current study may be combined with those from a previous study (NIDA protocol 417) which now reside in our repository protocol, 8002 and NIDA protocol 455.

Outcome measures- The primary outcome measures will be the difference in BOLD fMRI activation between drug-exposed participants and those without prenatal exposure to drugs of abuse.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants must be enrolled in the current UMB longitudinal study protocol.
  2. All participants will be between 14 and 20 years old (inclusive).
  3. All participants must be able to provide informed assent and have a parent/guardian who can provide informed consent or if 18 or older, be able to provide informed consent..

EXCLUSION CRITERIA:

1. Report of a history of significant medical/neurological illness that might interfere with imaging data such as HIV positive status, cerebral vascular accident (CVA), central nervous system (CNS) tumor, head trauma, multiple sclerosis (MS) or other demyelinating diseases, epilepsy, or movement disorders.
2. Metallic devices in the body that preclude MRI scanning, as determined by self and parent (guardian) report.
3. Current use of psychotropic medication that may alter attentional functioning (e.g., Clonidine, antipsychotics, Effexor, stimulants).
4. Currently using respiratory, cardiovascular, anticonvulsant or other medications that might interfere with the mechanisms producing the BOLD signal.
5. Pregnancy, which will be assessed by history during screening and by urine testing on scan days.
6. Claustrophobia by self and/or parent (guardian) report severe enough to preclude toleration of the scanning environment.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2011-05-15; Study Completion 2013-02-26

PRIMARY OUTCOMES:
The primary outcome measures will be the difference in BOLD fMRI activation between drug-exposed participants and those without prenatal exposure to drugs of abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Jo Salmeron, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- University of Maryland at Baltimore/MPRC, Catonsville, Maryland, United States

REFERENCES:
- [Background] Accornero VH, Morrow CE, Bandstra ES, Johnson AL, Anthony JC. Behavioral outcome of preschoolers exposed prenatally to cocaine: role of maternal behavioral health. J Pediatr Psychol. 2002 Apr-May;27(3):259-69. doi: 10.1093/jpepsy/27.3.259. PMID 11909933
- [Background] Bandstra ES, Morrow CE, Anthony JC, Accornero VH, Fried PA. Longitudinal investigation of task persistence and sustained attention in children with prenatal cocaine exposure. Neurotoxicol Teratol. 2001 Nov-Dec;23(6):545-59. doi: 10.1016/s0892-0362(01)00181-7. PMID 11792524
- [Background] Bandstra ES, Vogel AL, Morrow CE, Xue L, Anthony JC. Severity of prenatal cocaine exposure and child language functioning through age seven years: a longitudinal latent growth curve analysis. Subst Use Misuse. 2004 Jan;39(1):25-59. doi: 10.1081/ja-120027765. PMID 15002943